CLINICAL TRIAL: NCT05542160
Title: Effectiveness of IRK-19® on Body Weight Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Greenyn Biotechnology Co., Ltd. (Industry)
Collaborators: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: G-CAZ0040161110628-1
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Overweight; Metabolic Syndrome
MeSH Terms: conditions — Overweight; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Pumpkin seed extract (IRK-19)
- Treatment (Experimental): IRK-19 capsule
  Interventions: Dietary Supplement: Pumpkin seed extract (IRK-19)

INTERVENTIONS:
Dietary Supplement: Pumpkin seed extract (IRK-19) — Placebo: Dietary fiber powder, two capsules/day (600 mg/day), continued use for 3 months Treatment: Pumpkin seed extract powder, two capsules/day (600 mg/day), continued use for 3 months

SUMMARY:
This randomized, double-blind, placebo-controlled, and parallel clinical study aims to investigate the effectivness of a pumpkin seed extract (IRK-19®) on weight management.

ELIGIBILITY:
Inclusion Criteria:

1. BMI: 25-30 kg/m2
2. Waistline circumference: ˃ 80 cm

Exclusion Criteria:

1. Pregnant women or preparing for pregnancy.
2. Lactating women.
3. Women gave birth 6 months before the study.
4. Subject uses diuretic, corticosteroids, anti-depressant medications, or antipsychotic medications.
5. Subject has undertaken obesity-related surgeries within one year prior to the study or other surgeries within six months prior to the study.
6. Change of body weight of subject is over 5% within 3 months before the study.
7. Subject has serious diseases (e.g., cardiovascular diseases).
8. Cancer patient.
9. Subject has engaged in another study within 3 months before the study.
10. Subject uses another dietary supplement related to weight management during the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurement | Week 0
  Body weight
Anthropometric measurement | Week 6
  Body weight
Anthropometric measurement | Week 12
  Body weight
Anthropometric measurement | Week 0
  Waist circumference
Anthropometric measurement | Week 6
  Waist circumference
Anthropometric measurement | Week 12
  Waist circumference
Anthropometric measurement | Week 0
  Hip circumference
Anthropometric measurement | Week 6
  Hip circumference
Anthropometric measurement | Week 12
  Hip circumference
Body composition analysis | Week 0
  Body fat
Body composition analysis | Week 6
  Body fat
Body composition analysis | Week 12
  Body fat
Body composition analysis | Week 0
  Visceral fat
Body composition analysis | Week 6
  Visceral fat
Body composition analysis | Week 12
  Visceral fat
Body composition analysis | Week 0
  Subcutaneous fat
Body composition analysis | Week 6
  Subcutaneous fat
Body composition analysis | Week 12
  Subcutaneous fat
Biochemistry | Week 0
  Total cholesterol
Biochemistry | Week 6
  Total cholesterol
Biochemistry | Week 12
  Total cholesterol
Biochemistry | Week 0
  Triacylglycerol
Biochemistry | Week 6
  Triacylglycerol
Biochemistry | Week 12
  Triacylglycerol
Biochemistry | Week 0
  HDL
Biochemistry | Week 6
  HDL
Biochemistry | Week 12
  HDL
Biochemistry | Week 0
  LDL
Biochemistry | Week 6
  LDL
Biochemistry | Week 12
  LDL
Biochemistry | Week 0
  Adiponectin
Biochemistry | Week 6
  Adiponectin
Biochemistry | Week 12
  Adiponectin
Biochemistry | Week 0
  Lectin
Biochemistry | Week 6
  Lectin
Biochemistry | Weeks 12
  Lectin
Biochemistry | Week 0
  Fasting blood glucose
Biochemistry | Week 6
  Fasting blood glucose
Biochemistry | Week 12
  Fasting blood glucose
Biochemistry | Week 0
  Insulin
Biochemistry | Week 6
  Insulin
Biochemistry | Week 12
  Insulin

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Nung Lin, MD, Principal Investigator — WanFang Hospital
Locations (1):
- WanFang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No